CLINICAL TRIAL: NCT04237701
Title: Retrospective and Real-Time Monitoring of Heart Failure Across the Yale New Haven Health System Via a Live Registry
Brief Title: Real-Time Monitoring of Heart Failure Across the Yale New Haven Health System
Acronym: Yale-HF
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000026771; No NIH funding (Other: 10.11.23)
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction; Heart Failure With Preserved Ejection Fraction; Heart Failure NYHA Class IV
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Yale HF Registry is a live EHR based registry that allows for retrospective and real-time monitoring of Heart Failure case across the Yale New Haven Health System.

DETAILED DESCRIPTION:
Electronic Health Records based registries can be an important resource for precision medicine delivery by understanding the population burden of chronic diseases such as heart failure. These registries can allow for a deeper understanding of gaps in guideline recommended therapies among patients who are under the purview of large, integrated Therefore, we have created a live registry within the integrated Yale New Haven Health System-the Yale Heart Failure Registry-that includes all patients with a diagnosis of HF and has detailed information about demographics, comorbidities, laboratories, imaging, medications, and clinical outcomes (including hospital readmissions). The registry is updated daily and can be queried for clinically relevant questions aimed at quality improvement.

ELIGIBILITY:
Inclusion Criteria:

* Seen within the Yale New Haven Health System
* Diagnosis of heart failure

Exclusion Criteria:

* Age<18

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Retrospective and Real-Time Monitoring of Heart Failure Across the Yale New Haven Health System Via a Live Registry
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants hospitalized for heart failure | 10 years
  Heart Failure hospitalizations
Doses of therapies that comprise guideline directed medical therapy | 10 years
  Appropriate use of guideline recommended therapies. This will include doses of beta blockers, ACE inhibitors, ARBs, ARNI, SGLT2i, ICD use.

CONTACTS AND LOCATIONS:
Overall Officials: Nihar Desai, MD MPH, Study Director — Yale University; Tariq Ahmad, MD MPH, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Health System, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Data is on patients seen at Yale New Haven Health system and will be used for quality improvement.

REFERENCES:
- [Result] Greene SJ, Fonarow GC, DeVore AD, Sharma PP, Vaduganathan M, Albert NM, Duffy CI, Hill CL, McCague K, Patterson JH, Spertus JA, Thomas L, Williams FB, Hernandez AF, Butler J. Titration of Medical Therapy for Heart Failure With Reduced Ejection Fraction. J Am Coll Cardiol. 2019 May 21;73(19):2365-2383. doi: 10.1016/j.jacc.2019.02.015. Epub 2019 Mar 4. PMID 30844480
- [Derived] Ahmad T, Desai NR. Reimagining Evidence Generation for Heart Failure and the Role of Integrated Health Care Systems. Circ Cardiovasc Qual Outcomes. 2022 Apr;15(4):e008292. doi: 10.1161/CIRCOUTCOMES.121.008292. Epub 2022 Mar 11. No abstract available. PMID 35272506